CLINICAL TRIAL: NCT03063203
Title: An Open Label, Multicenter, Phase II Trial Testing Single Agent Decitabine in TP53 Mutated Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Single Agent Decitabine in TP53 Mutated Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Collaborators: Janssen Pharmaceuticals (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201911185-1001; 3P50CA171963-06S1 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-02-24 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia, Relapsed, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Decitabine (Experimental): * Cycle 1: All patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle
  * Cycle 2: Patients with bone marrow blast counts < 5% may receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of a 28-day cycle. All other patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle.
  * Cycle 3 and subsequent cycles: All patients will receive 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of the 28-day cycle
  Interventions: Drug: Decitabine; Procedure: Bone marrow biopsy/aspirate; Procedure: Peripheral blood draw; Procedure: Skin biopsy; Procedure: Buccal swab

INTERVENTIONS:
Drug: Decitabine — * After 2 cycles, patients with progressive disease or relapse (a clear progression with at least >20% bone marrow blasts and an increase of at least 50% from prior biopsy) should be removed from protocol and proceed to salvage treatment according to center preference
  * Transplant eligible patients who achieve CR, CRc, or CRi, after 3 cycles with a suitable donor will proceed to conditioning regimen and transplant
  * Transplant eligible patients with PR after 3 cycles may be removed from protocol and proceed to salvage treatment according to center preference
  * Transplant eligible patients with a suitable donor who achieve mLFS, CR, CRc, or CRi, may proceed to transplant after at 3 cycles
  * Transplant ineligible patients with (CR, CRc or CRi, PR) will continue on maintenance doses
  * Transplant ineligible patient with SD after cycle 4 may be removed from protocol and proceed to alternative treatment or continue on protocol according to treating physician's preference.
  Other Names: 5-aza-2'-deoxycytidine
Procedure: Bone marrow biopsy/aspirate — * Baseline, Cycle 1 Day 10, Cycle 1 Day 28, Cycle 2 Day 28, Cycle 3 Day 28, and Progression or relapse
  * Biopsy/aspirate on Cycle 1 Day 10 is for participants enrolled at Washington University only
  * Biopsy/aspirate on Cycle 2 Day 28 is at the discretion of the treating physician
Procedure: Peripheral blood draw — -Baseline, Cycle 1 Day 10, Cycle 1 Day 28, Cycle 2 Day 28, Cycle 3 Day 28, and Progression/Relapse
Procedure: Skin biopsy — * Optional but if refuse skin biopsy then participant can provided buccal swab
  * There is no required time frame for this sample - it may have been collected months or even years prior to the first dose of decitabine
  * If WBC at time of enrollment is >30,000/µl, skin biopsy should be collected at the time of C1D28 bone marrow biopsy or thereafter
Procedure: Buccal swab — -Baseline (if skin biopsy declined) and Cycle 2 Day 28

SUMMARY:
In this study, the investigators seek to determine whether decitabine therapy can improve outcomes, specifically overall survival this selected subset of acute myeloid leukemia (AML) patients with the poorest prognosis based on refractoriness to induction treatment and high risk genetic mutations.

ELIGIBILITY:
Inclusion Criteria:

* TP53 mutant AML. The presence of a TP53 mutation should be determined by Genoptix (or institutional preferred equivalent assay). Detection of a TP53 mutation at the time of initial diagnosis is sufficient for enrollment at the time of relapsed/refractory disease. Detection of a TP53 mutation in either the peripheral blood or bone marrow is adequate for enrollment. Alternatively, patients who have not had TP53 mutation analysis performed, but who have > 20% TP53 positive cells by immunohistochemistry detected on a bone marrow aspirate may also be enrolled,29 provided that mutation analysis is requested at the time of enrollment.
* Relapsed/refractory AML following 7+3 (or similar cytarabine containing induction chemotherapy for AML) disease detected by one of the following methods:

  * bone marrow blasts > 5%, or
  * Hematologics flow cytometry assay (threshold > 0.5%) (alternative equivalent assay may be substituted), or
  * Persistent cytogenetic abnormality (e.g. del5, del17p, etc), by FISH or conventional karotyping, or
  * Persistent TP53 mutation (at least 5 variant reads with at least 50x coverage) determined by Genoptix (or institutional preferred equivalent assay).
* Patients with > 10% blasts on a day +14 bone marrow biopsy following 7+3 may either be enrolled or may be treated with a course of standard re-induction (e.g. 5+2 or similar) and then re-evaluated for response. Eligible patients will meet any of the above criteria on a subsequent biopsy.
* Bone marrow and organ function as defined below:

  * Peripheral white blood cell count < 50,000/mcl (patients may receive hydroxyurea as necessary for cytoreduction),
  * Total bilirubin < 1.5 x upper limit of normal,
  * AST and ALT < 2.5 x upper limit of normal,
  * Serum creatinine < 2.0 x upper limit of normal, and,
* At least 18 years of age.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable
* Performance status ≤ 3

Exclusion Criteria:

* Prior treatment with either decitabine or azacitidine or an investigational agent
* Acute promyelocytic leukemia with PML-RARA or t(15;17).
* History of HIV, Hepatitis B, or Hepatitis C infection.
* Concurrent illness including, but not limited to, ongoing uncontrolled infection, symptomatic NYHA class 3 or 4 congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Radiation therapy within 14 days of enrollment.
* Chemotherapy administration in the 7 days preceding enrollment with the exception of hydroxyurea, which can be continued until Cycle 2. A washout period for oral tyrosine kinase inhibitors (e.g. Jakafi, etc) is not required, although tyrosine kinase inhibitors therapy must be discontinued prior to enrollment.
* Malignancies (other than AML) requiring active therapy or diagnosed within the last year, with the exception of non-melanoma skin cancer which can be treated or in situ malignancies (such as cervical, breast, prostate, etc.)
* Currently receiving any other investigational agents.
* Known central nervous system (CNS) leukemia or testicular involvement of leukemia
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or other agents used in the study.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test within 7 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Welch, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decitabine
Started | 17
Completed | 3
Not Completed | 14
Not completed — Chose alternative therapy | 3
Not completed — Death | 2
Not completed — Disease progression | 4
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 61 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Participants With TP53 Mutation
Description: * Overall survival (OS) is defined as the time from enrollment to death due to any cause. For a patient who is not known to be alive at the end of study follow up, observation of OS is censored on the date the patient was last known to be alive
  * To be evaluable for this outcome measure the participant would have to have received at least one dose of decitabine
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 17
days | 244 [116 to 390]

2. Secondary Outcome: Percentage of Responding TP53 Mutated Patients (CR, CRi)
Description: * Complete remission (CR) - Defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1,000/μL); platelet count >100 x 109/L (100,000/μL).
  * Complete remission with incomplete hematologic recovery (CRi): All CR criteria except for residual neutropenia - <1.0 x 109/L (1,000/μL) or thrombocytopenia -<100 x 109/L (100,000/μL)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine
Number analyzed (Participants) | 17
Participants | 5

3. Secondary Outcome: Time to Stem Cell Transplant Among Participants Who Are Suitable Candidates for Transplant and Have an Identified Donor
Description: * Document the number of days that it takes each participant to reach transplant
  * Transplant eligible participants are those who achieve complete remission (CR), cytogenetic complete remission (CRc), complete remission with incomplete hematologic recovery (CRi), or morphologic leukemia free state (mLFS) per 2017 ELN AML Recommendations.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 7
days | 117 [77 to 163]

4. Secondary Outcome: Median Time to Leukemia Relapse (TTLR) in Non-transplant Patients
Description: -Recurrence/morphologic relapse - Defined as relapse following complete remission is defined as reappearance of blasts in the blood or the finding of ≥ 5% blasts in the bone marrow, not attributable to any other cause. New dysplastic changes is considered relapse. If there are no blasts in the peripheral blood and 5-20% blasts in the bone marrow, bone marrow biopsy should be repeated in > 1 week to confirm relapse.
Time Frame: 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 4
days | 308 [64 to 374]

5. Secondary Outcome: Event-free Survival (EFS)
Description: -Event-free survival is defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, death due to any cause, or loss to follow up.
Time Frame: 2 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 17
days | 227 [64 to 354]

6. Secondary Outcome: Average Number of Hospital Days
Description: -Document number of hospital days that each participant stays and obtain average for all evaluable participants
Time Frame: During cycles 1 and 2 (60 days)
Measure: Mean (Full Range); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 17
days | 10.3 [2 to 28]

7. Secondary Outcome: Response Compared Between Patients With Morphologically Evident Disease Versus Patients With Molecularly Detected Disease at the Time of Enrollment
Description: * Morphologically evident disease (>5% blasts by cytomorphology)
  * Molecularly detected disease (disease detected with flow cytometry, cytogenetic, or mutational analysis if ≤ 5% blasts by cytomorphology)
  * Response will be assessed according to the 2017 European LeukemiaNet (ELN) Acute Myeloid Leukemia (AML) recommendations
Time Frame: Through 12 weeks
Population: Response was not evaluable for 2 patients with molecularly evident disease as their samples were hemodilute. Response was not evaluable for 1 patient with molecularly detected disease as their sample was hemodilute.
Measure: Count of Participants; unit: Participants
Groups:
- Morphologically Evident Disease; Molecularly Detected Disease: * Cycle 1: All patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle
  * Cycle 2: Patients with bone marrow blast counts < 5% may receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of a 28-day cycle. All other patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle.
  * Cycle 3 and subsequent cycles: All patients will receive 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of the 28-day cycle
Arm/Group | Morphologically Evident Disease | Molecularly Detected Disease
Number analyzed (Participants) | 6 | 8
Participants
  Complete remission with incomplete hematologic recovery (CRi) | 3 | 2
  Morphologic leukemia free state (mLFS) | 0 | 1
  Stable Disease (SD) | 2 | 4
  Progressive disease (PD) | 1 | 1

8. Secondary Outcome: Survival Compared Between Patients With Morphologically Evident Disease Versus Patients With Molecularly Detected Disease at the Time of Enrollment
Description: * Morphologically evident disease (>5% blasts by cytomorphology)
  * Molecularly detected disease (disease detected with flow cytometry, cytogenetic, or mutational analysis with ≤ 5% blasts by cytomorphology)
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Morphologically Evident Disease | Molecularly Detected Disease
Number analyzed (Participants) | 8 | 9
days | 215 [58 to 390] | 336 [61 to 557]

9. Secondary Outcome: Response Compared Between Patients With de Novo AML Versus Patients With Secondary AML Versus Patients With Treatment-related AML
Description: -Response will be assessed according to the 2017 European LeukemiaNet (ELN) Acute Myeloid Leukemia (AML) recommendations
Time Frame: Through 12 weeks
Population: 2 patients with de novo AML were not evaluable for this outcome measure because the samples were hemodilute. 1 patient with treatment related AML was not evaluable for this outcome measure because the samples were hemodilute.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With de Novo AML; Patients With Secondary AML; Patients With Treatment Related AML: * Cycle 1: All patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle
  * Cycle 2: Patients with bone marrow blast counts < 5% may receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of a 28-day cycle. All other patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle.
  * Cycle 3 and subsequent cycles: All patients will receive 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of the 28-day cycle
Arm/Group | Patients With de Novo AML | Patients With Secondary AML | Patients With Treatment Related AML
Number analyzed (Participants) | 6 | 2 | 6
Participants
  Complete remission with incomplete hematologic recovery (CRi) | 3 | 0 | 2
  Morphologic leukemia free state (mLFS) | 0 | 0 | 1
  Stable Disease (SD) | 3 | 1 | 2
  Progressive disease (PD) | 0 | 1 | 1

10. Secondary Outcome: Survival Compared Between Patients With de Novo AML Versus Patients With Secondary AML Versus Patients With Treatment-related AML
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Patients With de Novo AML | Patients With Secondary AML | Patients With Treatment Related AML
Number analyzed (Participants) | 8 | 2 | 7
days | 246 [106 to 557] | 235 [116 to 354] | 244 [58 to 454]

11. Secondary Outcome: Response Compared Between Patients With Presence of Cytogenetic Abnormalities in Addition to TP53 Mutations Versus Patients With Absence of Cytogenetic Abnormalities in Addition to TP53 Mutations
Description: as for outcome 9
Time Frame: 12 weeks
Population: Response was not evaluable for 3 patients with presence of cytogenetic abnormalities in addition to TP53 mutations as their response samples were hemodilute.
Measure: Count of Participants; unit: Participants
Groups:
- Presence of Cytogenetic Abnormalities in Addition to TP53 Mutations; Absence of Cytogenetic Abnormalities in Addition to TP53 Mutations: * Cycle 1: All patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle
  * Cycle 2: Patients with bone marrow blast counts < 5% may receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of a 28-day cycle. All other patients will receive decitabine 20 mg/m^2 IV infusion per day over one hour on Days 1-10 of a 28-day cycle.
  * Cycle 3 and subsequent cycles: All patients will receive 20 mg/m^2 IV infusion per day over one hour on Days 1-5 of the 28-day cycle
Arm/Group | Presence of Cytogenetic Abnormalities in Addition to TP53 Mutations | Absence of Cytogenetic Abnormalities in Addition to TP53 Mutations
Number analyzed (Participants) | 13 | 1
Participants
  Complete remission with incomplete hematologic recovery (CRi) | 5 | 0
  Morphologic leukemia free state (mLFS) | 1 | 0
  Stable Disease (SD) | 5 | 1
  Progressive disease (PD) | 2 | 0

12. Secondary Outcome: Survival Compared Between Patients With Presence of Cytogenetic Abnormalities in Addition to TP53 Mutations Versus Patients With Absence of Cytogenetic Abnormalities in Addition to TP53 Mutations
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Presence of Cytogenetic Abnormalities in Addition to TP53 Mutations | Absence of Cytogenetic Abnormalities in Addition to TP53 Mutations
Number analyzed (Participants) | 16 | 1
days | 254 [116 to 390] | NA [NA to NA] — The median survival with 95% confidence interval was not estimable due to an insufficient number of participants with events.

13. Secondary Outcome: Median Number of Hospital Stays
Description: -Document number of hospital days that each participant stays and obtain median for all evaluable participants
Time Frame: During cycles 1 and 2 (60 days)
Measure: Median (Full Range); unit: days
Arm/Group | Decitabine
Number analyzed (Participants) | 17
days | 9 [2 to 28]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until 30 days after last dose of therapy (may continue until time of transplantation or disease progression - estimated time of 3-6 months). All-cause mortality was collected from time of consent through completion of follow-up (for 2 years after last dose of decitabine or until the patient is lost to follow-up or dies).
Arm/Group | Decitabine
All-Cause Mortality (participants affected / at risk) | 15/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=17)
Bacteremia streptococcus (Infections and infestations) | 1
Facial cellulitis (Infections and infestations) | 1
Febrile neutropenia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=17)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Infections and infestations) | 4
Chest tightness (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Knots (General disorders) | 1
Injection site reaction (General disorders) | 2
Localized edema - right breast (General disorders) | 1
Chills (General disorders) | 3
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Infusion related reaction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cellulitis on shin (Infections and infestations) | 1
Staphylococcus epidermis (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 5
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 7
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Oily skin (Skin and subcutaneous tissue disorders) | 1
Traumatic fat necrosis (Skin and subcutaneous tissue disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03063203/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03063203/ICF_000.pdf